CLINICAL TRIAL: NCT06215391
Title: Customized Masks in Non-Invasive Mechanical Ventilation: An Innovative Approach Through 3D Printing
Brief Title: Customized Masks in Non-Invasive Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23/478
Record Dates: First submitted 2023-11-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: COPD, Severe Early-Onset; Ventilatory Failure; Als; Non Invasive Ventilation
Keywords: non invasive ventilation; 3d printed mask
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive, Severe Early-Onset; Hypoventilation; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Conceptual Hypothesis:
  The use of personalized 3D-printed masks may reduce leaks, adverse effects in the form of skin lesions, and the percentage of upper airway obstructive events in two distinct populations: patients with ALS and patients with COPD requiring inspiratory pressures greater than 22 cmH2O.
  Operational Hypothesis:
  The automatic AHI and the median leaks over 1 month are lower when the patient uses the custom-fit 3D-printed mask (M3D) compared to when they use the commercial mask (MC) that was prescribed.
  Statistical Hypothesis:
  H0: There are no differences in the median leaks over 1 month (and AHI) between commercial masks (MC) and personalized 3D-printed masks (M3D).
  H1: The median leaks are significantly lower during the month of using the personalized mask (M3D) than during the use of the commercial mask.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- commercial mask (No Intervention): Noninvasive ventilation delivered through a conventional mask as usual care
- 3d printed mask (Experimental): The customized mask will be obtained by merging the scanned surface with the base mask design using CAD 3D SolidWorks software, also available in the unit. In patients with edentulism, leak areas will be evaluated without dental prostheses.
  3D Printing
  Personalized oronasal masks will be manufactured following this procedure:
  * Design and manufacture of molds for each type of base mask and the personalized mold of the scanned surface, using stereolithography technology with suitable biocompatible resin such as BioMed Clear or White from FormLABS.
  * Manual injection of a biocompatible resin with a Shore A hardness of 18, such as SORTA-Clear™ 18, by joining the two molds. This Shore A hardness will provide appropriate elasticity for this type of mask, perfectly adapting to each patient's unique facial characteristics.
  Interventions: Device: 3d printed mask

INTERVENTIONS:
Device: 3d printed mask — * Concurrent, prospective, non-randomized inclusion, cross-over design. A minimum of 6 patients will be included for each group, COPD, and ALS.
  * T0: Patient enrollment (informed consent signing), retrospective review of the respirator log (1 month prior), variable extraction (extracting EDF files from the respirator log and data obtained from ResScan).
  * During the first week, a 3D scan of the patient's face will be conducted, and the personalized 3D-printed mask (M3D) will be manufactured.
  * Once ready, the mask will be fitted, and the 1-month evaluation period will begin (T1: after 1 month of M3D use). The respirator card will be downloaded in the same manner as at T0, and a respiratory polygraphy (RP) will be scheduled.
  * T2: At the end of the study month, the patient will resume using a similar MC, which is new and well-fitted. After one month of MC use, the respirator log will be reviewed, and a new RP will be conducted.
  Arms: 3d printed mask

SUMMARY:
In non-invasive mechanical ventilation (NIMV), the interface is the primary determinant of success, as adherence and quality of therapy mainly depend on it. The aim of this study is to investigate the usefulness of a customised mask approach to minimise leakage and upper airway obstruction. It will focus on ventilator registries and changes in the way they can be corrected with these customised masks.

The process involves 3D face scanning and dedicated computer-aided design. The processing and manufacturing of the masks is based on additive manufacturing through 3D printing.

DETAILED DESCRIPTION:
In non-invasive mechanical ventilation (NIMV), the interface is the primary determinant of success, as adherence and the quality of therapy depend mainly on it. A deteriorated or inadequate mask can lead to unintentional leaks or jaw and tongue displacements, thereby increasing obstructive events in the upper airway. There is a growing interest in the use of personalized masks designed using facial scanning and 3D printing technology. Previous studies have demonstrated their effectiveness in complex patients, such as premature neonates, and healthy individuals, successfully reducing leaks and skin sores.

The aim of the project is to demonstrate the utility of a 3D-printed, customised mask to improve the quality of ventilation, primarily by reducing leaks and mask-related obstructions in adult patients receiving home NIMV. Two usage periods of NIMV will be studied, one month with a personalized mask created through 3D printing (M3D) and another month with a commercial mask (MC). The primary variable under study will be the difference in leak levels between M3D and MC throughout the study month with each of them. Variables derived from respiratory polygraphy, performed with each mask, will also be included, in addition to the patient's experience.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled in the Home Mechanical Ventilation (HMV) program.
* Adherence of >4 hours per day.
* In the case of COPD, inspiratory pressures >18 cmH2O.
* Users of a Resmed HMV device to standardize and facilitate the analysis of the respirator log.
* Commercial masks (MC) in optimal condition, as assessed by the mechanical ventilation unit responsible during outpatient ventilation consultations.
* Presence of residual leaks (>5 LPM on average according to the respirator log - ResScan, unintentional leaks, with intentional leaks excluded by software).

Exclusion Criteria:

* Patients with tracheostomy or scheduled for tracheostomy.
* Patients on a waiting list for lung transplantation.
* Patients using HMV devices from manufacturers other than ResMed.
* Users who alternate between various MC models, where homogeneity in interface use cannot be assured.
* Refusal to provide consent.
* Patients with documented allergies to components of medical-grade silicone used in the production of M3D.
* Exacerbations requiring hospitalization or changes in medication or the respirator in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Modifications in leaks | 1 month
  Median daily leakage over the study month with each mask (MC and M3D), determined from the respirator log, extracted using ResScan® (Resmed®) software.

SECONDARY OUTCOMES:
Apnea Hypopnea Index | 1 month
  • Mean AHI over the study month with each mask, automatically recorded by the respirator software (ResScan®) for each mask period. IAH /AHI ranges from 0 to over 30 events per hour. A threshold of <10 is usually considered a sign of adequate ventilation. A minimal decrease of 20% will be considered clinically relevant
Comfort | 1 month
  • Patient comfort at the end of the one-month period with each mask (Likert scale). Likert scale ranges from Strongly uncomfortable to strongly comfortable
Adherence | 1 month
  • Adherence measured by the mean device usage (hours of use/days of use) and total days of use in 1 month (T0 vs. T1).
• Polygraphic variables | 1 month
  .1 Asynchrony Index

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitarios 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lujan M, Florez P, Pomares X. What Circuits, Masks and Filters Should Be Used in Home Non-Invasive Mechanical Ventilation. J Clin Med. 2023 Apr 4;12(7):2692. doi: 10.3390/jcm12072692. PMID 37048774

DOCUMENTS (1):
  • Informed Consent Form (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT06215391/ICF_000.pdf